CLINICAL TRIAL: NCT01079754
Title: The Comparison of 0.05 vs. 0.1 Milligram Spinal Morphine for Reducing Morphine Requirement After Vaginal Hysterectomy With/Without Anterior and Posterior Vaginoplasty
Brief Title: 0.05 Versus 0.1 mg Spinal Morphine for Reducing Morphine Requirement After Vaginal Hysterectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Sirilak Suksompong, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Si 073/2010
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Pain; Vaginal Hysterectomy
Keywords: Spinal morphine 0.05 mg; Spinal morphine
MeSH Terms: conditions — Pain | interventions — Analgesics, Opioid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spinal morphine 0.05 mg (Experimental): Patient received spinal morphine 0.05 mg
  Interventions: Drug: Spinal morphine 0.05 mg
- Spinal morphine 0.1 mg (Active Comparator): Patient received spinal morphine 0.1 mg
  Interventions: Drug: Spinal morphine 0.1 mg

INTERVENTIONS:
Drug: Spinal morphine 0.05 mg — Patient received spinal morphine 0.05 mg
  Other Names: opioids
  Arms: Spinal morphine 0.05 mg
Drug: Spinal morphine 0.1 mg — Patient received spinal morphine 0.1 mg
  Other Names: Opioids
  Arms: Spinal morphine 0.1 mg

SUMMARY:
This study aims to compare the efficacy of 0.05 mg and 0.1 mg spinal morphine in reducing postoperative morphine requirement in patients undergoing vaginal hysterectomy with/without anterior and posterior vaginoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Female ASA physical status 1-3
* Undergoing vaginal hysterectomy with/without anterior and posterior vaginoplasty
* Be able to operate patient-controlled analgesia (PCA)

Exclusion Criteria:

* Allergy to the study drugs
* History of bleeding tendency
* Infection at the back
* Refuse to spinal anesthesia
* History of CAD or CVA

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The total amount of morphine that the patient required during the first 24-h postoperative. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Suksompong, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of medicine, Siriraj Hospital, Bangkok, Thailand